CLINICAL TRIAL: NCT04622839
Title: Post-Operative Pain Control Following Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Shoulder and Elbow Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00248454
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-04

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Diclofenac

STUDY DESIGN:
Intervention Model Description: Participants undergoing shoulder surgery will be randomized into one of the three study arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants will be masked to the aspect of post-operative pain management being manipulated in this study; investigator and outcomes assessor will be masked to randomization (group assignment) of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will not be aware of the relation to the group they are randomized into in comparison to the other study groups; for example, if they were assigned a higher or lower frequency of ice usage (with Intervention 1 being frequency of ice usage), etc.
  Interventions: Other: Tylenol and NSAIDS (Ibuprofen, diclofenac)
- Group 2 (Experimental): Participants will not be aware of the relation to the group they are randomized into in comparison to the other study groups; for example, if they were assigned a higher or lower frequency of ice usage (with Intervention 1 being frequency of ice usage), etc.
  Interventions: Other: Tylenol and NSAIDS (Ibuprofen, diclofenac)
- Group 3 (Experimental): Participants will not be aware of the relation to the group they are randomized into in comparison to the other study groups; for example, if they were assigned a higher or lower frequency of ice usage (with Intervention 1 being frequency of ice usage), etc.
  Interventions: Other: Tylenol and NSAIDS (Ibuprofen, diclofenac)

INTERVENTIONS:
Other: Tylenol and NSAIDS (Ibuprofen, diclofenac) — This study will assess an aspect of perioperative care relating to pain control. Subjects will not be aware of which aspect is randomized, but will be given a list of possible aspects which will include the intervention (listed below):
  * Agents used in nerve block (lidocaine vs ropivacaine)
  * Location of injection for analgesic
  * Use of over-the-counter pain management (including but not limited to acetaminophen, ibuprofen, naproxen, etc.)
  * Type of initial opioid prescribed (including but not limited to oxycodone, tramadol, hydrocodone, etc.)
  * Number of pills in the initial opioid prescription
  * Instructions for sling wear (duration of use or type of sling)
  * Ice usage (duration of use and frequency of use)
  Blinding the participant to the randomized aspect of this study will help prevent bias in patient responses for outcome scores and medication usage.

SUMMARY:
This study will evaluate overall opioid and non-narcotic analgesic use following surgical treatment for shoulder pathology, and recommend evidence based guidelines for standardized postoperative pain management.

DETAILED DESCRIPTION:
There is currently very limited information in the literature regarding postoperative pain medication consumption following orthopedic shoulder surgery. To fill this knowledge gap, this study will evaluate overall opioid consumption in morphine milligram equivalents following surgical treatment for shoulder pathology.

ELIGIBILITY:
Inclusion Criteria:

* Opioid-naive adults age 18-90 years old planning to undergo surgical treatment for shoulder pathology with the PI at Johns Hopkins Shoulder Service (Columbia, Odenton clinic sites; Howard County General Hospital/Johns Hopkins Hospital operative sites) will be included.

Exclusion Criteria:

* Patients with prior history of opioid misuse, addiction, or chronic pain
* Patients taking chronic pain medication or have taken opioid medication in the past 3 months will be excluded due to risk of developing drug tolerances that could affect the amount of pain medication consumed after surgery An exception will be made for those who have used narcotic medication for fracture-related events, and expect to undergo surgical treatment for fracture repair (ORIF or arthroplasty)
* Patients with BMI < 18.5 or > 39.9
* Patients with a history of adverse reaction and/or allergy to oxycodone
* Patients lacking the ability to consent will also be excluded.
* Patients whose primary residence is outside the United States will be excluded.
* Patients who are unable to complete questionnaires due to medical condition, psychiatric illness, or significant language barrier will also be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Morphine milligram equivalents (MMEs) consumed | 2 weeks postop
  Total possible narcotic pain medication use in MME's
Opioid Prescription Refills | 2 weeks postop
  number and quantity of opioid prescription refills
Office Contacts | 2 weeks postop
  Number of times patient contacted the office via telephone, MyChart, or email

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) score | 2-4 months postop
  standardized questionnaire for the assessment of shoulder function; single score which ranges from 0-100 with higher score reflecting higher function

CONTACTS AND LOCATIONS:
Overall Officials: Umasuthan Srikumaran, M.D., Principal Investigator — Johns Hopkins Orthopedics
Locations (1):
- Howard County General Hospital, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: No